CLINICAL TRIAL: NCT01667081
Title: A Long-Term Follow-Up Study to Evaluate the Durability of Virologic Response and/or Viral Resistance Patterns of Subjects With Chronic Hepatitis C Who Have Been Previously Treated With MK-5172 in a Prior Clinical Trial
Brief Title: Durability of Virologic Response and/or Viral Resistance Patterns in Participants With Chronic Hepatitis C Who Have Been Previously Treated With Grazoprevir (MK-5172) (MK-5172-017)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 5172-017; 2012-002232-85 (EudraCT Number)
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected and retained for purposes of Deoxyribonucleic acid (DNA) testing and plasma will be retained for future biomedical research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Grazoprevir: Participants who previously received grazoprevir as study treatment on a prior study.
  Interventions: Drug: Grazoprevir

INTERVENTIONS:
Drug: Grazoprevir — Participants previously received study treatment with grazoprevir at the dose and frequency specified in the study protocol. Grazoprevir was not administered to participants in the course of this follow-up study.

SUMMARY:
This is a three-year (except for participants with chronic kidney disease [CKD] or cirrhosis) multicenter study to follow participants who received at least one dose of grazoprevir (MK-5172) in a previous study to determine whether they remain hepatitis C virus (HCV)-Ribonucleic acid (RNA) negative over time, and to determine if they have developed antiviral resistance. The study will also evaluate long-term adverse events in this population. Participants from MK-5172-052 (NCT02092350) with CKD or cirrhosis will be followed for five years.

DETAILED DESCRIPTION:
As of Amendment 03, the study design is revised such that continued enrollment will only be for participants who failed prior therapy with a grazoprevir regimen. Participants with CKD enrolled from MK-5172-052 (NCT02092350) will continue enrollment regardless of prior treatment-response and remain in this study for five years, while participants enrolled from all other studies with HCV RNA less than the lower limit of quantitation (LLOQ) will be discontinued and end their participation after the next scheduled visit. In addition, participants who receive other HCV treatments concurrent with this follow-up study or received other HCV treatments prior to this study will be discontinued and their data excluded from analysis.

As of Amendment 04, the protocol has been updated to include enrollment of pediatric participants from protocol MK-5172-079 (NCT03379506). Enrollment is limited to participants who experienced virologic failure associated with 1 or more treatment-emergent resistant associated substitutions (RASs) present at 12 weeks after receiving grazoprevir treatment in prior treatment study MK-5172-079 (NCT03379506).

ELIGIBILITY:
Inclusion Criteria:

* Previously participated in a HCV treatment protocol that included grazoprevir in the treatment regimen
* Must enroll in the present study within three months of the last study visit of their previous protocol in which they received a grazoprevir-containing regimen
* For Amendment 03: Adult participants must have received a grazoprevir-containing regimen in a prior trial and have been identified as having failed therapy in that study
* For Amendment 04: Pediatric participants must have received at least 1 dose of a grazoprevir-containing regimen and experienced virologic failure with 1 or more associated treatment-emergent RASs at Follow-up Week 12 in MK-5172-079 (NCT03379506)

Exclusion Criteria:

* Has received HCV therapy after completion of the protocol-defined grazoprevir treatment trial regimen and before or after entry into this follow-up study
* For Amendment 03: Has failed therapy due to re-infection, defined as an HCV RNA sample with a different genotype than the baseline genotype in the prior treatment study, or an HCV RNA sample determined to be reinfection by phylogenetic analysis with comparison to the baseline sequence in the prior treatment study
* For Amendment 03: Has failed therapy and received retreatment with HCV therapy, except in the case where they were re-treated in a Merck-sponsored protocol

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric participants previously treated with a grazoprevir-containing regimen while enrolled in a Merck study. All participants enrolled having failed therapy from prior studies (except MK-5172-052 [NCT02092350]) will be followed for 3 years in the current follow-up study, and all participants enrolled from MK-5172-052 (irrespective of prior response) will be followed for 5 years in the current follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 2438 (Actual)
Dates: Start 2012-10-17 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Lahser F, Galloway A, Hwang P, Palcza J, Brunhofer J, Wahl J, Robertson M, Barr E, Black T, Asante-Appiah E, Haber B. Interim analysis of a 3-year follow-up study of NS5A and NS3 resistance-associated substitutions after treatment with grazoprevir-containing regimens in participants with chronic HCV infection. Antivir Ther. 2018;23(7):593-603. doi: 10.3851/IMP3253. Epub 2018 Jul 24. PMID 30038064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2438 adult Hepatitis C Virus (HCV)-infected participants who were previously treated in 18 prior clinical trials, enrolled in this study.
Pre-assignment Details: Of the 2438 participants, three participants were excluded from all analyses. Two participants enrolled in error failed to receive at least 1 dose of Grazoprevir (GZR) in a prior study (each received a comparator regimen in a prior base study) and 1 participant had insufficient long-term follow-up data (participant withdrew consent on Day 27).
Groups:
- Grazoprevir (GZR) 100 mg + Elbasvir (EBR) 50 mg +/- Ribavirin (RBV): Participants previously received GZR 100mg +EBR 50mg with or without RBV in a prior study.
- Other GZR Regimen: Participants previously received at least one dose of GZR in a prior study
Period: Overall Study
Arm/Group | Grazoprevir (GZR) 100 mg + Elbasvir (EBR) 50 mg +/- Ribavirin (RBV) | Other GZR Regimen
Started | 1909 | 526
Completed | 132 | 169
Not Completed | 1777 | 357
Not completed — Death | 43 | 3
Not completed — Lost to Follow-up | 99 | 48
Not completed — Physician Decision | 16 | 2
Not completed — Participants were discontinued due to amendment 3 which modified the study discontinuation criteria | 1529 | 269
Not completed — Withdrawal by Subject | 90 | 35

BASELINE CHARACTERISTICS:
Groups:
- GZR 100 mg + EBR 50 mg +/- RBV: Participants previously received GZR 100mg +EBR 50mg with or without RBV in a prior study.
- Total: Total of all reporting groups
Arm/Group | GZR 100 mg + EBR 50 mg +/- RBV | Other GZR Regimen | Total
Number analyzed (Participants) | 1909 | 526 | 2435
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (11.0) | 49.7 (11.4) | 51.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 785 | 238 | 1023
  Male | 1124 | 288 | 1412
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 135 | 68 | 203
  Not Hispanic or Latino | 1730 | 444 | 2174
  Unknown or Not Reported | 44 | 14 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 283 | 12 | 295
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 253 | 35 | 288
  White | 1345 | 470 | 1815
  More than one race | 21 | 6 | 27
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Viral Relapse
Description: Viral relapse is defined as any participant who has confirmed HCV Ribonucleic acid (RNA) ≥ Lower limit of quantification (LLoQ) of 15 IU/mL and had achieved sustained virologic response (SVR) in the follow up in the prior treatment study. Time to relapse is defined as the time from last dose of study therapy taken in the prior treatment study until the date where HCV RNA is ≥LLoQ.
Time Frame: Up to ~60 months after enrollment in this study
Population: All participants who achieved SVR during the follow-up period of the prior treatment study and did not start any new HCV therapy between the end of the prior treatment study and entry in this study
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | GZR 100 mg + EBR 50 mg +/- RBV | Other GZR Regimen
Number analyzed (Participants) | 1837 | 495
Months | NA [NA to NA] — Median time to viral relapse and interquartile range not reached due to the low rate of late virologic relapse. | NA [NA to NA] — Median time to viral relapse and interquartile range not reached due to the low rate of late virologic relapse.

2. Primary Outcome: Persistence of Treatment-Emergent Nonstructural Protein (NS)3 and NS5A Resistance-associated Substitutions (RASs) in Participants With HCV Genotype (GT) 1a Infections
Description: In adult participants with HCV RNA ≥1000 IU/mL at entry or during the study period, HCV sequence analysis was performed to evaluate the presence of RASs and the persistence of RASs over time.
Time Frame: Up to ~60 months after enrollment in this study
Population: Participants met the criteria of virologic failure either in the prior base study or had HCV RNA Target detected, quantifiable [TD(q)] at entry in current study. Participants did not receive new HCV therapy between the end of the prior base study and entry into this study. Only HCV genotype infections that had adequate reference information were included.
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR +/- RBV: NS3 RASs: Participants previously received EBR and GZR with or without RBV in a prior study and had treatment-emergent NS3 RASs
- EBR/GZR +/- RBV: NS5A RASs: Participants previously received EBR and GZR with or without RBV in a prior study and had treatment-emergent NS5A RASs
- EBR/GZR +/-RBV: Both NS3 and NS5A RASs: Participants previously received EBR and GZR with or without RBV in a prior study and had both treatment-emergent NS3 and NS5A RASs
- GZR + Pegylated Interferon/Ribavirin (PR): NS3 RASs: Participants previously received GZR and PR for 12 weeks in a prior study and had treatment-emergent NS3 RASs
Arm/Group | EBR/GZR +/- RBV: NS3 RASs | EBR/GZR +/- RBV: NS5A RASs | EBR/GZR +/-RBV: Both NS3 and NS5A RASs | GZR + Pegylated Interferon/Ribavirin (PR): NS3 RASs
Number analyzed (Participants) | 31 | 31 | 31 | 16
Participants
  Failure | 22 | 25 | 18 | 11
  24 weeks post failure | 10 | 25 | 8 | 2
  48 weeks post failure: number analyzed (Participants) | 30 | 30 | 30 | 16
  48 weeks post failure | 6 | 22 | 4 | 2
  96 weeks post failure: number analyzed (Participants) | 21 | 21 | 21 | 15
  96 weeks post failure | 4 | 15 | 3 | 1
  ≥144 weeks post failure: number analyzed (Participants) | 17 | 17 | 17 | 8
  ≥144 weeks post failure | 2 | 11 | 1 | 1

3. Primary Outcome: Persistence of Treatment-Emergent NS3 and NS5A RASs in Participants With HCV Genotype 1b Infections
Description: as for outcome 2
Time Frame: Up to ~60 months after enrollment in this study
Population: Participants met the criteria of virologic failure either in the prior base study or had HCV RNA TD(q) at entry in current study. Participants did not receive new HCV therapy between the end of the prior base study and entry into this study. Only HCV genotype infections that had adequate reference information were included.
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR+/- RBV: NS3 RASs: Participants previously received EBR and GZR with or without RBV in a prior study and had treatment-emergent NS3 RASs
- EBR/GZR +/-RVB: Both NS3 and NS5A RASs: Participants previously received EBR and GZR with or without RBV in a prior study and had both treatment-emergent NS3 and NS5A RASs
- GZR + RBV or PR: NS3 RASs: Participants previously received GZR and RBV or PR for 12 weeks in a prior study and had treatment-emergent NS3 RASs
Arm/Group | EBR/GZR+/- RBV: NS3 RASs | EBR/GZR +/- RBV: NS5A RASs | EBR/GZR +/-RVB: Both NS3 and NS5A RASs | GZR + RBV or PR: NS3 RASs
Number analyzed (Participants) | 9 | 9 | 9 | 5
Participants
  Failure | 4 | 7 | 2 | 3
  24 weeks post failure | 2 | 7 | 0 | 1
  48 weeks post failure: number analyzed (Participants) | 6 | 6 | 6 | 4
  48 weeks post failure | 1 | 5 | 0 | 1
  96 weeks post failure: number analyzed (Participants) | 4 | 4 | 4 | 4
  96 weeks post failure | 1 | 3 | 0 | 1
  ≥144 weeks post failure: number analyzed (Participants) | 3 | 3 | 3 | 4
  ≥144 weeks post failure | 0 | 3 | 0 | 1

4. Primary Outcome: Persistence of Treatment-Emergent NS3 and NS5A RASs in Participants With Genotype 4 Infections
Description: as for outcome 2
Time Frame: Up to ~60 months after enrollment in this study
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR: NS3 RASs: Participants previously received EBR and GZR in a prior study and had treatment-emergent NS3 RASs
- EBR/GZR: NS5A RASs: Participants previously received EBR and GZR in a prior study and had treatment-emergent NS5A RASs
- EBR/GZR: Both NS3 and NS5A RASs: Participants previously received EBR and GZR in a prior study and had both treatment-emergent NS3 and NS5A RASs
Arm/Group | EBR/GZR: NS3 RASs | EBR/GZR: NS5A RASs | EBR/GZR: Both NS3 and NS5A RASs
Number analyzed (Participants) | 5 | 5 | 5
Participants
  Failure | 2 | 4 | 2
  24 weeks post failure | 1 | 3 | 1
  48 weeks post failure | 1 | 2 | 1
  96 weeks post failure | 1 | 2 | 1
  ≥144 weeks post failure | 1 | 2 | 1

5. Primary Outcome: Number of Participants Who Experienced a Drug-Related Adverse Event (AE) During the Long-Term Follow-Up
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The study investigator determined whether the adverse event was drug-related.
Time Frame: Up to ~ 60 months after enrollment in this study
Population: All participants treated with GZR in a prior study. Three participants were excluded from analysis; two participants enrolled in error failed to receive at least one dose of GZR in a prior study (each received a comparator regimen in a prior base study) and one participant had insufficient long-term follow-up data (participant withdrew consent on Day 27).
Measure: Count of Participants; unit: Participants
Arm/Group | GZR 100 mg + EBR 50 mg +/- RBV | Other GZR Regimen
Number analyzed (Participants) | 1909 | 526
Participants | 1 | 1

6. Primary Outcome: Number of Participants Who Experienced a Drug-Related Serious Adverse Event (SAE) During the Long-Term Follow-Up
Description: A serious adverse event (SAE) is any adverse experience occurring at any dose that either results in death, is life threatening, results in a persistent or significant disability/incapacity, results in or prolongs an existing inpatient hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose (whether accidental or intentional), or other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse experience when, based upon appropriate medical judgment, the event may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed previously. The study investigator determined whether the adverse event was drug-related.
Time Frame: Up to ~60 months after enrollment in this study
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GZR 100 mg + EBR 50 mg +/- RBV | Other GZR Regimen
Number analyzed (Participants) | 1909 | 526
Participants | 1 | 1

7. Primary Outcome: Number of Participants Who Experienced an Event of Clinical Interest (ECI) During the Long-Term Follow-Up
Description: An ECI includes spontaneous bacterial peritonitis, variceal bleeding, ascites, encephalopathy, hepatorenal syndrome, hepatocellular carcinoma, liver transplant, cardiovascular disease limited to angina and myocardial infarction, neurologic disorders limited to transient ischemic attack (TIA) or stroke, graft rejection in participants who have undergone liver or kidney transplant, or one of the following in participants from the MK-5172-052 (NCT02092350) base study: kidney transplant, decreased estimated glomerular filtration rate (eGFR), new onset diabetes, cryoglobulinemia, or post transplantation glomerulonephritis.
Time Frame: Up to ~60 months after enrollment in this study
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GZR 100 mg + EBR 50 mg +/- RBV | Other GZR Regimen
Number analyzed (Participants) | 1909 | 526
Participants | 98 | 4

ADVERSE EVENTS:
Time Frame: From first visit in follow-up (Screening/Baseline) up to ~60 months after enrollment in this study
Description: The all-cause mortality population includes all enrolled participants (N=2438). The serious adverse events and other adverse events population excludes three enrolled participants- two enrolled in error who received a comparator regimen in a prior base study and one participant had insufficient long-term follow up data (participant withdrew consent on day 27).
Groups:
- Non-GZR Regimen: Participants received a non-GZR regimen in a prior study
Arm/Group | GZR 100 mg + EBR 50 mg +/- RBV | Other GZR Regimen | Non-GZR Regimen
All-Cause Mortality (participants affected / at risk) | 44/1909 | 3/527 | 0/2
Serious Adverse Events (participants affected / at risk) | 100/1909 | 4/526 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1909 | 0/526 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GZR 100 mg + EBR 50 mg +/- RBV (N=1909) | Other GZR Regimen (N=526) | Non-GZR Regimen (N=0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0) | NA
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | NA
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | NA
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | NA
Cardiac arrest (Cardiac disorders) | 4 (4) | 0 (0) | NA
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | NA
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | NA
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | NA
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0) | NA
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | NA
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Chest pain (General disorders) | 1 (2) | 0 (0) | NA
Death (General disorders) | 8 (8) | 0 (0) | NA
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | NA
Sudden death (General disorders) | 1 (1) | 0 (0) | NA
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | NA
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | NA
Kidney transplant rejection (Immune system disorders) | 1 (1) | 0 (0) | NA
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | NA
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | NA
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | NA
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | NA
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | NA
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | NA
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Glomerular filtration rate decreased (Investigations) | 5 (5) | 0 (0) | NA
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 1 (1) | NA
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | NA
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
Cerebrovascular accident (Nervous system disorders) | 2 (3) | 0 (0) | NA
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | NA
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | NA
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | NA
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | NA
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | NA
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1) | NA
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | NA
Transient ischaemic attack (Nervous system disorders) | 3 (5) | 0 (0) | NA
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | NA
Chronic kidney disease (Renal and urinary disorders) | 7 (7) | 0 (0) | NA
End stage renal disease (Renal and urinary disorders) | 17 (17) | 0 (0) | NA
Glomerulonephritis chronic (Renal and urinary disorders) | 2 (2) | 0 (0) | NA
Renal failure (Renal and urinary disorders) | 6 (6) | 0 (0) | NA
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0) | NA
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT01667081/Prot_SAP_000.pdf